CLINICAL TRIAL: NCT04428970
Title: Intracranial Pressure Monitoring Following Traumatic Brain Injury - Evaluation of Indications, Complications, and Significance of Follow-up Imaging.
Brief Title: Intracranial Pressure (ICP) Monitoring Following Traumatic Brain Injury (TBI)
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Haider, M.D., Ph.D., Medical University of Vienna
Other Study IDs: 2086/2019
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Traumatic Brain Injury
Keywords: Intracranial pressure monitoring
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TBI patients with ICP monitoring: Patients with severe TBI (GCS<9 on arrival) receiving invasive ICP monitoring
  Interventions: Procedure: Invasive ICP monitoring

INTERVENTIONS:
Procedure: Invasive ICP monitoring — Insertion of a parenchymal pressure measuring probe

SUMMARY:
The aim of this retrospective cohort study is to evaluate complications rates, indications, and the utility of follow-up imaging studies of ICP measurement in severe TBI patients.

ELIGIBILITY:
Inclusion Criteria:

* Severe Traumatic Brain Injury (GCS<9 on arrival)
* Implantation of invasive intracranial parenchymal ICP monitoring

Exclusion Criteria:

* incomplete data records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients transferred to our department after severe TBI who had received invasive ICP monitoring will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Complications | up to 30 days
  Intervention-related complications

SECONDARY OUTCOMES:
Clinical outcome | up to 30 days
  Outcome at discharge measured by the Glasgow Outcome Scale (GOS), range 1(death) - 5 (good recovery)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Universtiy of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No